CLINICAL TRIAL: NCT02169752
Title: Ambrisentan for the Improvement in Right Ventricular Strain in Scleroderma Associated Pulmonary Arterial Hypertension
Acronym: AMERICA-PAH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left National Jewish Health
Sponsor: National Jewish Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS-2716
Record Dates: First submitted 2014-05-06; First posted 2014-06-23 (Estimated); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Pre-Pulmonary Atrial Hypertension
Keywords: Pre-Pulmonary Atrial Hypertension
MeSH Terms: interventions — ambrisentan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ambrisentan (Active Comparator): Subjects will be randomly assigned in a 1:1 ration according to the computer generated random numbers to receive either placebo (sugar pill) or ambrisentan.
  Interventions: Drug: Ambrisentan
- Placebo (Placebo Comparator): Subjects will be randomly assigned in a 1:1 ration according to the computer generated random numbers to receive either placebo (sugar pill) or ambrisentan.
  Interventions: Drug: Ambrisentan

INTERVENTIONS:
Drug: Ambrisentan — Subjects will be randomized 1:1 ratio according to computer generated random numbers to receive either "placebo" or ambrisentan 5mg daily for one month followed by 10 mg daily for the 5 months in a double-blinded manner.
  Other Names: Letairis

SUMMARY:
This research study is looking at the use of the drug ambrisentan and if it can improve right ventricle function in people with systemic sclerosis-associated pre-pulmonary arterial hypertension. It is also looking at using right ventricle function changes as a marker of disease severity.

DETAILED DESCRIPTION:
This research study is looking at the use of the drug ambrisentan and if it can improve right ventricle function in people with systemic sclerosis-associated pre-pulmonary arterial hypertension. It is also looking at using right ventricle function changes as a marker of disease severity.

Pre-pulmonary arterial hypertension is a borderline elevation in blood pressure in the lungs. Pre-pulmonary arterial hypertension is not currently treated with the drug therapies that are used for pulmonary arterial hypertension. It represents a group of patients that are at risk for developing pulmonary arterial hypertension.

The administration of ambrisentan is the experimental part of this study. Ambrisentan has not been approved by the FDA for use of improving right ventricle function in people with pre-pulmonary arterial hypertension. You will still receive your normal clinical care.

The purpose of this study is to learn more about ambrisentan and its role in treating systemic sclerosis-associated pre-pulmonary arterial hypertension. Ambrisentan is already approved for use in people with systemic sclerosis-associated pulmonary arterial hypertension, but this study wants to research its role in people with pre-pulmonary arterial hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years, < 80 years
* Systemic sclerosis with any of the following features:

  1. Duration of Raynaud's phenomena >8 years
  2. Anticentromere antibody positivity
  3. isolated nucleolar-pattern ANA positivity
  4. Extensive telangiectasias
  5. DLCO < 60% in the absence of extensive ILD
  6. FVC%/DLCO% >1.6
  7. Unexplained dyspnea
* Right heart catheterization-proven pre PAH (mean PAP 20-25 mmHg and pulmonary capillary wedge pressure <15 mmHg)
* Systolic blood pressure >100 mmHg
* Reliable contraception for women of childbearing age
* Informed consent

Exclusion Criteria:

* < 18 years or > 80 years
* Left ventricular ejection fraction < 55%
* Systolic or diastolic left ventricular congestive heart failure
* Liver disease (abnormal AST/ALT, chronic hepatitis, or cirrhosis)
* Extensive ILD or FVC< 60%
* Pregnant
* Breast-feeding women
* Cyclosporine use

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-09; Primary Completion 2017-05-25 (Actual); Study Completion 2017-05-25 (Actual)

PRIMARY OUTCOMES:
Improvement in right ventricular (RV) myocardio strain > 2% | 1, 3 and 6 months
  Assess for tolerance, gas exchange, and therapeutic benefit, resting oximetry, six minute walk with oximetry, pulmonary function testing with diffusion capacity (DLCO), and functional class will be assessed prior to ambrisentan initiation, and 1,3, and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Brett Fenster, MD, Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Health, Denver, Colorado, United States